CLINICAL TRIAL: NCT04752046
Title: Is the Maxillectomy Patient's Quality of Life Affected by Palatal Defect Reconstruction Via Scapular Free Flab or Obturator? A Randomized Clinical Trial
Brief Title: Scapular Flap Versus Obturator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofaciall surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Maxillary Defect Reconstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obturator group (Active Comparator): patients with resected maxillary defects were managed with surgical obturator
  Interventions: Procedure: maxillary cancer resection
- scapular flap group (Active Comparator)
  Interventions: Procedure: maxillary cancer resection

INTERVENTIONS:
Procedure: maxillary cancer resection — patient with maxillary cancer will resected and reconstructed

SUMMARY:
The aim of this study was to evaluate and compare quality of life (QoL) outcomes of scapular island flap versus maxillary obturator reconstruction after partial maxillectomy. patients indicated for maxillectomy were allocated randomly to two equal-sized groups. Control group patients underwent reconstruction with a surgical obturator, while intervention group patients underwent scapular island flap reconstruction

ELIGIBILITY:
Inclusion Criteria:

* n0 lymph node
* older than 18ys

Exclusion Criteria:

* patients who recived radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
patient quality of life | 6month
  patient quality of life will evaluated with byversion 4 of UW-QOL

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt